CLINICAL TRIAL: NCT00300547
Title: Preoperative Assessment for Synchronous Carcinoma or Polyps With MR Colonography in Patients With Obstructing Cancer. A Prospective Study.
Brief Title: Preoperative Assessment for Synchronous Carcinoma or Polyps With Magnetic Resonance (MR) Colonography
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Herlev Hospital (Other)
Collaborators: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Michael Achiam, MD, Herlev Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KA05030-MA; KA05030
Record Dates: First submitted 2006-03-08; First posted 2006-03-09 (Estimated); Last update posted 2010-08-18 (Estimated); Status verified 2006-03

CONDITIONS: Obstructing Colorectal Cancer
Keywords: colorectal cancer; polyps; Virtual colonoscopy; synchronous carcinoma; MR colonography
MeSH Terms: conditions — Colorectal Neoplasms; Polyps

INTERVENTIONS:
Procedure: MR colonography — Altered planned surgical procedure if MR colonoscopy reveals synchronous cancer or larger polyps

SUMMARY:
The purpose of this study is to diagnose possible synchronous carcinomas and polyps with magnetic resonance (MR) colonography in patients booked for operation because of carcinoma in the descending or sigmoid colon, where a preoperative full colonoscopy is not possible. Two days before colonography, patients ingest a 200 ml Barium sulfate solution four times a day, which will render fecal masses "invisible" on the following MR colonography. The study is primarily a feasibility study with altered operative strategy as a secondary end-point. Gold standard is colonoscopy and operation.

ELIGIBILITY:
Inclusion Criteria:

* Obstructing colorectal cancer

Exclusion Criteria:

* Suspicion of IBD
* Pacemaker
* Metal in the body
* Claustrophobia
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-03; Primary Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Feasibility of MR colonography to diagnose possible synchronous carcinomas and polyps | 3

SECONDARY OUTCOMES:
Altered operative strategy due to findings on MR colonography | 3

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Achiam, MD, Principal Investigator — Department of Radiology Copenhagen University Hospital Herlev
Locations (1):
- Department of Radiology Copenhagen University Hospital Herlev, Copenhagen, Denmark